CLINICAL TRIAL: NCT02143726
Title: Randomized Phase II Study of Sorafenib With or Without Everolimus in Patients With Radioactive Iodine Refractory Hurthle Cell Thyroid Cancer
Brief Title: Sorafenib Tosylate With or Without Everolimus in Treating Patients With Advanced, Radioactive Iodine Refractory Hurthle Cell Thyroid Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A091302; U10CA180821 (NIH); NCI-2014-00623 (Registry Identifier: NCI Clinical Trials Reporting Office)
Record Dates: First submitted 2014-05-19; First posted 2014-05-21 (Estimated); Results first posted 2022-04-04 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-01

CONDITIONS: Refractory Hurthle Cell Thyroid Cancer
MeSH Terms: conditions — Thyroid cancer, Hurthle cell | interventions — Sorafenib; Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- sorafenib (Active Comparator): Patients receive sorafenib 400 mg PO twice daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients with progressive disease may cross over and receive everolimus 10 mg PO once daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: sorafenib
- sorafenib and everolimus (Experimental): Patients receive sorafenib 400 mg PO twice daily and everolimus 5 mg PO once daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: sorafenib; Drug: everolimus

INTERVENTIONS:
Drug: sorafenib — Given PO
  Other Names: Nexavar ®, BAY 43-9006
Drug: everolimus — Given PO
  Other Names: RAD001, Afinitor ®
  Arms: sorafenib and everolimus

SUMMARY:
This randomized phase II trial studies the effects, good and bad, of using everolimus along with sorafenib tosylate versus sorafenib tosylate alone in treating patients with advanced radioactive iodine refractory thyroid cancer. Sorafenib tosylate and everolimus may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. The addition of everolimus to sorafenib tosylate may cause more shrinkage of thyroid cancer and may prevent it from growing but it could also cause more side effects than sorafenib tosylate alone. It is not yet known whether this treatment with sorafenib tosylate and everolimus is better, the same, or worse than sorafenib tosylate alone.

DETAILED DESCRIPTION:
This randomized Phase II trial will compare the progression-free survival (PFS) of sorafenib and everolimus versus sorafenib alone in patients with radioactive iodine refractory hurthle cell thyroid cancer. Prior studies have shown that the median PFS is generally around 4.5 months for sorafenib alone in this disease population. It is hoped that the combination of everolimus and sorafenib can increase the median PFS to at least 9 months. In addition to PFS, this trial will also compare the confirmed response rate, overall survival (OS) and adverse event rates between sorafenib and everolimus vs. sorafenib alone. The primary and secondary objectives for the study are listed below.

Primary Objective:

To compare the progression free survival between sorafenib and everolimus versus sorafenib alone in patients with radioactive iodine refractory Hurthle cell thyroid cancer

Secondary Objective:

To compare the confirmed response rate, overall survival and adverse event rates between sorafenib and everolimus versus sorafenib alone.

Treatment will continue until disease progression or unacceptable adverse events. Patients will be followed for 5 years after randomization.

ELIGIBILITY:
Eligibility Criteria:

1. Central pathology review submission - Patients must have 10 representative hematoxylin and eosin (H&E) stained thyroid tissue slides OR tumor block available for submission to central pathology review. This review is mandatory prior to registration to confirm eligibility.
2. Measurable disease - Patients must have measurable disease by Response Evaluation Criteria In Solid Tumors (RECIST) criteria, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as ≥ 20 mm with conventional techniques or as ≥ 10 mm with spiral computed tomography (CT) scan. CT must be performed within 28 days of registration.
3. Radioactive iodine (RAI) - refractory disease defined as 1 or more of the following:

   * Patients who have received greater than 600 mCi of radioactive iodine in their lifetime OR
   * RAI-avid metastatic lesion which remained stable in size or progressed despite RAI treatment within 9 months of RAI treatment OR
   * 10% or more increase in serum thyroglobulin (on thyroid-stimulating hormone [TSH]-suppression) within 9 months of RAI treatment OR
   * Index metastatic lesion non-RAI avid on a diagnostic RAI scan OR
   * Presence of fluorodeoxyglucose (FDG) avid metastatic lesions on positron emission tomography (PET)/CT scan (standardized uptake values [SUV]max > 5 of any single lesion)
4. Progressive disease defined by RECIST criteria ≤ 14 months
5. Patients must have metastatic disease or locally advanced unresectable disease
6. Prior treatment

   * Patients may have received prior radiation therapy to index lesions ≥ 28 days prior to registration on this protocol if there has been documented progression by RECIST criteria. Prior radiation therapy to the non-index lesions is allowed if ≥ 28 days prior to registration on this protocol.
   * Prior RAI therapy is allowed if ≥ 90 days prior to registration on this protocol and evidence of progression (as defined above) has been documented in the interim (a diagnostic study using < 10 mCi of RAI is not considered RAI therapy).
   * Prior chemotherapy is allowed if ≥ 28 days prior to registration on this protocol.
   * Patient may have received any number of prior lines of therapy.
   * No prior use of sorafenib or an mammalian target of rapamycin (mTOR) (including phosphoinositide 3-kinase [PI3k] or protein kinase B [AKT]) inhibitor for the treatment of thyroid cancer.
7. No history of major surgery ≤ 28 days of registration
8. No history of intracranial brain metastasis
9. Cardiovascular disease. No history of any of the following ≤ 6 months of registration:

   * Myocardial infarction or unstable angina
   * New York Heart Association grade III or greater congestive heart failure
   * Cerebrovascular accident
   * Grade 3 or 4 peripheral ischemia
   * Grade 3 or 4 thromboembolic event
10. Liver disease: No history of the following:

    * Child Pugh Class B or C liver disease
    * "Chronic active" hepatitis defined as:

      1. Hepatitis B surface antigen (HBsAg) > 6 months
      2. Serum hepatitis B virus (HBV) deoxyribonucleic acid (DNA) 20,000 IU/ml (105 copies/ml), lower values 2,000-20,000 IU/ml (104-105 copies/ml) are often seen in hepatitis B e antigen (HBeAg)-negative chronic hepatitis B
      3. Persistent or intermittent elevation in alanine aminotransferase (ALT)/aspartate aminotransferase (AST) levels
      4. Liver biopsy showing chronic hepatitis with moderate or severe necroinﬂammation
11. No history of gastrointestinal fistula or gastrointestinal perforation < 90 days of registration.
12. No known history of prolonged QT syndrome
13. No Grade 3 or 4 hypertension (systolic blood pressure [BP] >160 and or diastolic BP > 100) that cannot be controlled with medication prior to registration.
14. Concomitant medications:

    * Chronic concomitant treatment with strong inhibitors of cytochrome P450 3A4 (CYP3A4) is not allowed on this study. Patients on strong CYP3A4 inhibitors must discontinue the drug for 14 days prior to registration on the study.
    * Chronic concomitant treatment with strong CYP3A4 inducers is not allowed. Patients must discontinue the drug 14 days prior to the start of study treatment.
    * Patients requiring anticoagulation must be on stable dose of medication prior to registration.
15. Not pregnant and not nursing, because this study involves an investigational agent whose genotoxic, mutagenic and teratogenic effects on the developing fetus and newborn are unknown. Therefore, for women of childbearing potential only, a negative serum pregnancy test done ≤ 7 days prior to registration is required.
16. Age ≥ 18 years
17. Eastern Cooperative Oncology Group (ECOG) Performance Status ≤ 2
18. Required Initial Laboratory Values:

    * Absolute neutrophil count (ANC) ≥ 1,500/mm^3
    * Platelet count ≥ 100,000/mm^3
    * Creatinine ≤ 1.5 mg/dL OR
    * Calculated creatinine clearance ≥ 30 mL/min
    * Total bilirubin ≤ 1.5 x upper limits of normal (ULN)
    * Serum glutamic oxaloacetic transaminase (SGOT) (AST) ≤ 2.5 x ULN
    * Fasting serum cholesterol ≤ 300 mg/dL
19. Documentation of disease: Histologic Documentation - Eligible patients must have histopathologically confirmed Hürthle cell thyroid cancer by central review.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2014-10-09 (Actual); Primary Completion 2021-01-28 (Actual); Study Completion 2028-08-06 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Sherman, M.D., Study Chair — Memorial Sloan Kettering Cancer Center
Locations (21):
- United States (21):
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Northwestern University, Chicago, Illinois
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Sleepy Hollow, Sleepy Hollow, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - Southeastern Medical Oncology Center-Clinton, Clinton, North Carolina
  - Southeastern Medical Oncology Center-Goldsboro, Goldsboro, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Southeastern Medical Oncology Center-Jacksonville, Jacksonville, North Carolina
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Mercy Health System, Janesville, Wisconsin

REFERENCES:
- [Derived] Matsuura D, Yuan A, Wang L, Ranganath R, Adilbay D, Harries V, Patel S, Tuttle M, Xu B, Ghossein R, Ganly I. Follicular and Hurthle Cell Carcinoma: Comparison of Clinicopathological Features and Clinical Outcomes. Thyroid. 2022 Mar;32(3):245-254. doi: 10.1089/thy.2021.0424. PMID 35078345

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1 (Sorafenib): Patients receive sorafenib 400 mg PO twice daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients with progressive disease may cross over and receive everolimus 10 mg PO once daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
- Arm 2 (Sorafenib and Everolimus): Patients receive sorafenib 400 mg PO twice daily and everolimus 5 mg PO once daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Arm 1 (Sorafenib) | Arm 2 (Sorafenib and Everolimus)
Started | 18 | 17
Received Everolimus After Disease Progression | 11 | 0
Completed | 16 | 17
Not Completed | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 (Sorafenib) | Arm 2 (Sorafenib and Everolimus) | Total
Number analyzed (Participants) | 16 | 17 | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.4 (13.4) | 65.6 (7.4) | 65.5 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 2 | 8
  Male | 10 | 15 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 14 | 16 | 30
  Unknown or Not Reported | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 12 | 15 | 27
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival
Description: Progression Free Survival (PFS) was defined as the time from randomization to the first of either disease progression or death from any cause. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: 4 years and 4 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm 1 (Sorafenib) | Arm 2 (Sorafenib and Everolimus)
Number analyzed (Participants) | 16 | 17
Months | 9.4 [5.5 to NA] — Upper limit not reached due to insufficient number of participants with events | 24.7 [6.1 to 33.8]
Statistical Analysis 1: Comparison: Arm 1 (Sorafenib) vs Arm 2 (Sorafenib and Everolimus); Test type: Superiority; p = 0.0918, Log Rank; Stratified 1-sided log-rank test (stratified by ECOG performance status, prior systemic treatment for hürthle thyroid cancer, and treating site); Hazard Ratio (HR) = 0.56, 95% CI 2-sided [0.23 to 1.33]

2. Secondary Outcome: Confirmed Response Rate
Description: A patient will be classified as a confirmed response per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: 4 years 4 months
Measure: Number; unit: Proportion of participants
Arm/Group | Arm 1 (Sorafenib) | Arm 2 (Sorafenib and Everolimus)
Number analyzed (Participants) | 16 | 17
Proportion of participants | 0.188 | 0.235

3. Secondary Outcome: Overall Survival
Time Frame: 5 years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm 1 (Sorafenib) | Arm 2 (Sorafenib and Everolimus)
Number analyzed (Participants) | 16 | 17
Months | NA [25.7 to NA] — Median and Upper limit not reached due to insufficient number of participants with events | 40.1 [38.2 to NA] — Upper limit not reached due to insufficient number of participants with events
Statistical Analysis 1: Comparison: Arm 1 (Sorafenib) vs Arm 2 (Sorafenib and Everolimus); Test type: Superiority; p = 0.3976, Log Rank; Hazard Ratio (HR) = 1.62, 95% CI 2-sided [0.53 to 4.96]

4. Secondary Outcome: Number of Participants With Grade 3 or Higher Adverse Events
Description: The maximum grade for each type of adverse event will be summarized using CTCAE version 4.0. The frequency and percentage of grade 3+ adverse events will be compared between the 2 treatment arms.
Time Frame: 4 years 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 (Sorafenib) | Arm 2 (Sorafenib and Everolimus)
Number analyzed (Participants) | 16 | 17
Participants | 10 | 12

ADVERSE EVENTS:
Time Frame: 4 years 3 months
Arm/Group | Arm 1 (Sorafenib) | Arm 2 (Sorafenib and Everolimus)
All-Cause Mortality (participants affected / at risk) | 5/17 | 8/17
Serious Adverse Events (participants affected / at risk) | 10/17 | 6/17
Other Adverse Events (participants affected / at risk) | 17/17 | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (Sorafenib) (N=17) | Arm 2 (Sorafenib and Everolimus) (N=17)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Eye disorders - Other, specify (Eye disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0)
Gen disord and admin site conds-Oth spec (General disorders) | 1 (1) | 0 (0)
Gallbladder infection (Infections and infestations) | 1 (1) | 0 (0)
Kidney infection (Infections and infestations) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 1 (1)
Tracheal obstruction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (1)
Weight loss (Investigations) | 2 (5) | 0 (0)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Stroke (Nervous system disorders) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Surgical and medical proced - Oth spec (Surgical and medical procedures) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (Sorafenib) (N=17) | Arm 2 (Sorafenib and Everolimus) (N=17)
Anemia (Blood and lymphatic system disorders) | 13 (86) | 15 (165)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac disorders - Other, specify (Cardiac disorders) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1) | 2 (2)
Cataract (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (2)
Bloating (Gastrointestinal disorders) | 1 (2) | 1 (2)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (2)
Diarrhea (Gastrointestinal disorders) | 13 (160) | 15 (140)
Dry mouth (Gastrointestinal disorders) | 2 (2) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 2 (3)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (2)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (2)
Mucositis oral (Gastrointestinal disorders) | 4 (5) | 2 (7)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (10)
Edema limbs (General disorders) | 1 (6) | 2 (3)
Facial pain (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 15 (207) | 15 (222)
Fever (General disorders) | 1 (1) | 0 (0)
Gen disord and admin site conds-Oth spec (General disorders) | 1 (1) | 1 (1)
Pain (General disorders) | 4 (9) | 2 (3)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Infections and infestations - Oth spec (Infections and infestations) | 1 (1) | 1 (1)
Injury to carotid artery (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (2) | 1 (1)
Alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0)
Cholesterol high (Investigations) | 1 (6) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 3 (9)
Neutrophil count decreased (Investigations) | 4 (12) | 2 (3)
Platelet count decreased (Investigations) | 10 (86) | 7 (46)
Weight loss (Investigations) | 14 (133) | 13 (156)
Anorexia (Metabolism and nutrition disorders) | 1 (2) | 3 (10)
Hyperglycemia (Metabolism and nutrition disorders) | 13 (176) | 14 (131)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 2 (6) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (12) | 2 (7)
Neck pain (Musculoskeletal and connective tissue disorders) | 3 (4) | 1 (2)
Cognitive disturbance (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (2)
Dysgeusia (Nervous system disorders) | 2 (5) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Muscle weakness left-sided (Nervous system disorders) | 0 (0) | 1 (1)
Paresthesia (Nervous system disorders) | 0 (0) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 1 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 2 (4)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Renal calculi (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 2 (4) | 2 (3)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary tract pain (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary urgency (Renal and urinary disorders) | 1 (1) | 1 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (4) | 2 (5)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (5)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (10) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (5)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Palmar-plantar erythrodysesthesia syndrm (Skin and subcutaneous tissue disorders) | 12 (113) | 12 (94)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (5) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (3) | 7 (22)
Skin and subcut tissue disord - Oth spec (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Surgical and medical proced - Oth spec (Surgical and medical procedures) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 15 (233) | 16 (266)
Thromboembolic event (Vascular disorders) | 0 (0) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-11): https://cdn.clinicaltrials.gov/large-docs/26/NCT02143726/Prot_SAP_000.pdf